CLINICAL TRIAL: NCT00494702
Title: Achievement of a Targeted Saturation in Extremely Low Gestational Age Neonates Resuscitated With Low or High Oxygen Concentration: A Prospective Randomized Trial
Brief Title: Oxygen Toxicity in the Resuscitation in Extremely Premature Infants
Acronym: OXTOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion Para La Investigacion Hospital La Fe (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: INSTITUTO DE SALUD CARLOS III -MINISTERIO DE SANIDAD Y CONSUMO -SPAIN, MAXIMO VENTO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIO51O5; FISPI05105
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Birth Asphyxia; Premature Birth
Keywords: Asphyxia; Resuscitation; Oxidative stress; Prematurity; Follow up
MeSH Terms: conditions — Asphyxia Neonatorum; Premature Birth; Asphyxia | interventions — Resuscitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LOX (Experimental): Low saturation group of premature infants that will be kept within preset limits of 85-89%
  Interventions: Procedure: Resuscitation
- HOX (Active Comparator): HOX group of premature infants will be kept within preset saturation limits of 90-93%
  Interventions: Procedure: Resuscitation

INTERVENTIONS:
Procedure: Resuscitation — Use of inspiratory fraction of oxygen needed to achieve oxygen saturation in the preset limits 85-88%
  Arms: LOX
Procedure: Resuscitation — Oxygen inspiratory fraction needed to keep oxygen saturation in the preset limits of 90-93%
  Arms: HOX

SUMMARY:
The investigators hypothesize that using low oxygen concentrations during resuscitation of extremely premature infants will avoid oxidative stress derived damage and improve outcome.

DETAILED DESCRIPTION:
This is a prospective randomized trial enrolling premature infants of less than 28 weeks gestation. Patients are randomly assigned to become resuscitation with an initial oxygen inspiratory fraction (FiO2) of 30% or 90%. Main objective is to reach a target saturation of 85% at 15 min of life.

Immediately after birth pre-and-postductal pulse oximeters are set and oxygen saturation (SpO2) continuously monitored and registered as long as the patient requires oxygen supplementation. FiO2 is stepwise adjusted (increased or decreased 10%) every 90 sec according to heart rate, SpO2 and responsiveness.

Blood samples are drawn from umbilical cord and at day 1, 2 and 7 from peripheral vein to determine oxidative stress markers (GSH, GSSG), angiogenic factors (VEGF, VEGF receptors, Angiopoietin), pro-inflammatory markers (IL8, TNF alfa) and pro-apoptotic markers (Fas Ligand; Cytochrome C).

Urine is collected every day during the first week of life to determine oxidative stress markers (8-oxo-dG; O-tyrosine; F2 isoprostanes; Isofurans).

Babies are followed in the NICU and clinical condition recorded. Serial examinations for ROP and Auditory evoked potentials will be performed. Neurodevelopmental outcome is evaluated at 2 years of postnatal life. Main outcome: Achievement of a target saturation of 85% at 15 min of life. Secondary outcomes: acute complications during delivery; chronic complications (BPD, ROP, IPVH); mortality in the neonatal period.

ELIGIBILITY:
Inclusion Criteria:

* Prematurity of less than 28 weeks gestation

Exclusion Criteria:

* Severe malformations
* Chromosomopathies
* Informed consent not signed

Ages: 1 Minute to 3 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2005-04; Primary Completion 2008-03 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Achievement of a targeted saturation of 85% at 15 min of life. | 30 min

SECONDARY OUTCOMES:
Neonatal mortality | 28 days of life
Oxidative stress | at day 1, 2 and 7
Bronchopulmonary dysplasia | 36 weeks postconceptional age
Retinopathy of prematurity | 40 weeks postconceptional
Neurodevelopment | 24 months postnatal

CONTACTS AND LOCATIONS:
Overall Officials: Maximo Vento, Phd, Md, Principal Investigator — Hospital Universitario La Fe
Locations (1):
- Servicio de Neonatologia, Valencia, Valencia, Spain

REFERENCES:
- [Background] Vento M, Asensi M, Sastre J, Garcia-Sala F, Pallardo FV, Vina J. Resuscitation with room air instead of 100% oxygen prevents oxidative stress in moderately asphyxiated term neonates. Pediatrics. 2001 Apr;107(4):642-7. doi: 10.1542/peds.107.4.642. PMID 11335737
- [Background] Vento M, Asensi M, Sastre J, Lloret A, Garcia-Sala F, Minana JB, Vina J. Hyperoxemia caused by resuscitation with pure oxygen may alter intracellular redox status by increasing oxidized glutathione in asphyxiated newly born infants. Semin Perinatol. 2002 Dec;26(6):406-10. doi: 10.1053/sper.2002.37312. PMID 12537311
- [Background] Vento M, Asensi M, Sastre J, Lloret A, Garcia-Sala F, Vina J. Oxidative stress in asphyxiated term infants resuscitated with 100% oxygen. J Pediatr. 2003 Mar;142(3):240-6. doi: 10.1067/mpd.2003.91. PMID 12640369
- [Background] Saugstad OD, Ramji S, Irani SF, El-Meneza S, Hernandez EA, Vento M, Talvik T, Solberg R, Rootwelt T, Aalen OO. Resuscitation of newborn infants with 21% or 100% oxygen: follow-up at 18 to 24 months. Pediatrics. 2003 Aug;112(2):296-300. doi: 10.1542/peds.112.2.296. PMID 12897277
- [Background] Saugstad OD, Ramji S, Vento M. Resuscitation of depressed newborn infants with ambient air or pure oxygen: a meta-analysis. Biol Neonate. 2005;87(1):27-34. doi: 10.1159/000080950. Epub 2004 Sep 20. PMID 15452400
- [Background] Vento M, Sastre J, Asensi MA, Vina J. Room-air resuscitation causes less damage to heart and kidney than 100% oxygen. Am J Respir Crit Care Med. 2005 Dec 1;172(11):1393-8. doi: 10.1164/rccm.200412-1740OC. Epub 2005 Sep 1. PMID 16141440
- [Background] Saugstad OD, Ramji S, Vento M. Oxygen for newborn resuscitation: how much is enough? Pediatrics. 2006 Aug;118(2):789-92. doi: 10.1542/peds.2006-0832. No abstract available. PMID 16882835
- [Background] Bookatz GB, Mayer CA, Wilson CG, Vento M, Gelfand SL, Haxhiu MA, Martin RJ. Effect of supplemental oxygen on reinitiation of breathing after neonatal resuscitation in rat pups. Pediatr Res. 2007 Jun;61(6):698-702. doi: 10.1203/pdr.0b013e3180534171. PMID 17426659
- [Derived] Escrig R, Arruza L, Izquierdo I, Villar G, Saenz P, Gimeno A, Moro M, Vento M. Achievement of targeted saturation values in extremely low gestational age neonates resuscitated with low or high oxygen concentrations: a prospective, randomized trial. Pediatrics. 2008 May;121(5):875-81. doi: 10.1542/peds.2007-1984. PMID 18450889